CLINICAL TRIAL: NCT04633395
Title: Treating Pregnancy Related Insomnia With Music: a Randomised Control Trial
Brief Title: Treating Pregnancy Related Insomnia With Music
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Caregiving+
Record Dates: First submitted 2020-11-03; First posted 2020-11-18 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy Related; Sleep Disturbance; Insomnia
Keywords: Music; Sleep; Insomnia; Non-pharmaceutic; Sleep disturbances
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Pregnant women in the third trimester will be randomised to 2 different groups (intervention group, and active control group).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music before bedtime (Experimental): Participants will be listening to music before bedtime for a duration of up to 1 hour each night, in a total treatment period of 4 weeks. Participants will also receive the sleep hygiene guidelines, and be told to follow these.
  Interventions: Other: Music; Behavioral: Sleep hygiene
- Sleep hygiene (Active Comparator): Participants will be given sleep hygiene guidelines, and be asked to follow these during the total treatment period of 4 weeks.
  Interventions: Behavioral: Sleep hygiene

INTERVENTIONS:
Other: Music — The participant can choose between 5 different soothing playlists
  Arms: Music before bedtime
Behavioral: Sleep hygiene — These are behavioural guidelines to help establish a better sleep pattern

SUMMARY:
This study aims to examine the effects of 4 weeks music listening at bedtime on sleep quality during the third trimester of pregnancy.

DETAILED DESCRIPTION:
50-60% of pregnant women suffer from insomnia during pregnancy. Pregnancy-related insomnia is often neglected due to a lack of suitable and safe treatments. This study aims to evaluate the effectiveness of music compared to sleep hygiene on sleep quality in a population of first-time pregnant women in the final stages of pregnancy. A post pregnancy follow-up will be completed to test if potential effects of the treatment might last into early motherhood (1-3 months postpartum).

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 years or above, pregnant non-mothers
* Have a sufficient level of Danish (verbal) to understand and respond to the questions and task instructions
* Pregnant women will be enrolled in gestation week 29.

Exclusion Criteria:

* Postnatal depression, i.e. a score of 12 or above on the EPDS questionnaire
* Comorbid psychiatric disorder (i.e. epilepsy and depression)
* Using sleep medication
* Working more than two night shifts per week
* History of sleep disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Sleep quality | Change from baseline to the end of the 4-week intervention, (post-treatment data will be collected immediately after completion of intervention). Furthermore, between group differences at follow up, up to 3 months postpartum
  Pittsburgh Sleep Quality Index. Scoring from 0-21 with higher numbers meaning more severe sleep problems. Cut-off score at 5.
Sleep quality - insomnia symptoms | Change from baseline to the end of the 4-week intervention, (post-treatment data will be collected immediately after completion of intervention). Furthermore, between group differences at follow up, up to 3 months postpartum
  Insomnia Severity Index. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).

SECONDARY OUTCOMES:
Depressive symptoms | Change from baseline to the end of the 4-week intervention, (post-treatment data will be collected immediately after completion of intervention). Furthermore, between group differences at follow up, up to 3 months postpartum
  Edinburgh Postnatal Depression Scale. Maximum score of 30, and minimum of 0. The higher the score, the more severe the symptoms. A Danish cut-off score at 11 is used.
Stress | Change from baseline to the end of the 4-week intervention, (post-treatment data will be collected immediately after completion of intervention). Furthermore, between group differences at follow up, up to 3 months postpartum
  Perceived Stress Scale. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Pre-sleep arousal | Change from baseline to the end of the 4-week intervention, (post-treatment data will be collected immediately after completion of intervention). Furthermore, between group differences at follow up, up to 3 months postpartum
  The Pre-Sleep Arousal Scale (PSAS) contains 16 items with eight symptoms of cognitive (e.g., intrusive thoughts) and eight symptoms of somatic (e.g., sweating) arousal experienced at bed- time. A total score from 8 to 40 is computed for both subscales with higher scores indicating higher arousal.
Prenatal attachment | Change from baseline to the end of the 4-week intervention, (post-treatment data will be collected immediately after completion of intervention). Furthermore, between group differences at follow up, up to 3 months postpartum
  Prenatal attachment Inventory. It consists of 21 Likert-type items with a 4-point response scale (1 = almost never, 2 = sometimes, 3 = often, 4 = almost always). Total scores can range from 21 to 84, with high scores indicating higher levels of prenatal attachment.
Anxiety | Change from baseline to the end of the 4-week intervention, (post-treatment data will be collected immediately after completion of intervention). Furthermore, between group differences at follow up, up to 3 months postpartum
  State- Trait Anxiety Inventory. It consists of two subtests - trait and state anxiety. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety.
Postpartum bonding | Between group differences at follow up, up to 3 months postpartum
  Postpartum Bonding Questionnaire. The PBQ consists of 25 statements about mothers' feelings, where mothers answer how well the statement applies to them on a six-point scales ranging from 0 to 5, with higher values indicating more problems. Min. score: 0, Max score: 125
Childbirth experience | Between group differences at follow up, up to 3 months postpartum
  Childbirth Experience Questionnaire. For 19 of the items the response format is a 4-point Likert Scale whereas the last three items use a visual analogue scale (VAS). The scoring range is 1 to 4 where higher ratings reflect more positive experiences. Min = 22. Max = 88

OTHER OUTCOMES:
Sleep apnea | Pre- and post treatment (at the end date of the 4 week intervention) measurements to ensure the participant has not developed sleep apnea
  Epworth Sleepiness Scale. 8 items scored from 0-3. Interpretation: 0-5 lower normal daytime sleepiness. 6-10 normal daytime sleepiness. 11-12 mild excessive daytime symptoms. 13-15 moderate excessive daytime symptoms. 16-24 severe excessive daytime symptoms.
Music reward | Baseline measurement only.
  Barcelona Music Reward Questionnaire. The BMRQ is a 20-item questionnaire that examines five main facets that characterize musical reward experience in individuals: musical seeking, emotion evocation, mood regulation, social reward and sensory-motor. Participants indicate the level of agreement with each statement by using a five-point scale ranging from "fully disagree" (1) to "fully agree" (5). The contribution of each facet to the overall music reward experience is quantified by a numerical value obtained upon completion of the survey. A score for global sensitivity to music reward is also provided, which was obtained as the weighted sum of participants' scores (i.e., factor score). The mean value of each factor is 50, and the standard deviation is 10. Standard values are therefore located between 40 and 60. Punctuations below 40 indicate low values in this particular facet, whereas values above 60 indicate high values (the same applies to the global sensitivity to music reward)

CONTACTS AND LOCATIONS:
Overall Officials: Morten L Kringelbach, Professor, Principal Investigator — Aarhus University anf University of Oxford
Locations (1):
- Center for Music In the Brain, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoegholt NF, Kraenge CE, Vuust P, Kringelbach M, Jespersen KV. Music and Sleep Hygiene Interventions for Pregnancy-Related Insomnia: An Online Randomized Controlled Trial. J Midwifery Womens Health. 2025 May-Jun;70(3):387-395. doi: 10.1111/jmwh.13699. Epub 2024 Oct 17. PMID 39417384
- [Derived] Jespersen KV, Pando-Naude V, Koenig J, Jennum P, Vuust P. Listening to music for insomnia in adults. Cochrane Database Syst Rev. 2022 Aug 24;8(8):CD010459. doi: 10.1002/14651858.CD010459.pub3. PMID 36000763